CLINICAL TRIAL: NCT03465046
Title: Modified Constraint Induced Movement Therapy and Bimanual Intensive Therapy in Children With Hemiplegia. Comparative Study
Brief Title: Intensive Therapies in Children With Hemiplegia
Acronym: CIMT/BIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Palomo Carrión, physiotherapist, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nº11, thesis SDDB USAL
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Infantile Hemiplegia
Keywords: infantile hemiplegia; upper extremity; physical therapy
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low performance group 1 (Experimental): Protocol 1 will be the intervention administered with 80 h modified constraint induced movement therapy and 20 h bimanual intensive therapy
  Interventions: Combination Product: intensive therapies(CIMT/BIT): protocol 1 or protocol 2
- low performance group 2 (Experimental): Protocol 2 will be the intervention administered with 80h bimanual intensive therapy and 20h modified constraint induced movement therapy
  Interventions: Combination Product: intensive therapies(CIMT/BIT): protocol 1 or protocol 2
- moderate-high performance group1 (Experimental): Protocol 1 will be the intervention administered with 80 h modified constraint induced movement therapy and 20 h bimanual intensive therapy
  Interventions: Combination Product: intensive therapies(CIMT/BIT): protocol 1 or protocol 2
- moderate-high performance group 2 (Experimental): Protocol 2 will be the intervention administered with 80h bimanual intensive therapy and 20h modified constraint induced movement therapy
  Interventions: Combination Product: intensive therapies(CIMT/BIT): protocol 1 or protocol 2

INTERVENTIONS:
Combination Product: intensive therapies(CIMT/BIT): protocol 1 or protocol 2 — The therapies applied in both protocols are intensive therapies that allow the execution of unimanual activities or bimanual activities with the affected upper limb with different doses.
  the protocols were carried out at home through the family

SUMMARY:
This is a comparative study where two protocols of intensive therapies will be applied to study the improvements in the functional performance of the affected upper limb of children with hemiparesis and check whether to increase their quality of life.

DETAILED DESCRIPTION:
the intervention protocols combine different doses of intensive therapy, being 80 hours of modified constraint induced movement therapy followed by 20 hours for protocol 1 and protocol 2 would be the application of protocol 1 inverted, with this, the investigators want to compare how both protocols interfere in the function of the affected upper limb of children with different levels of bimanual functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Unilateral Infantile Cerebral Palsy, Congenital Infantile Hemiparesis.
* Ages between 5 to 10 years.
* Levels of I-III within the , manual ability classification system, MACS.
* Levels of I-III within the gross motor function classification system, GMFCS

Exclusion Criteria:

- Diseases not associated with infantile hemiparesis.

* Low cognitive level to understand the execution of activities.
* Surgeries of the upper extremity during the 6 months prior to the intervention.
* Structured contractures in the affected upper extremity that cause functional impotence.
* Botulinum toxin two months prior to the intervention and application of it during the treatment.
* Epilepsy not controlled pharmacologically

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
bimanual functional performance, "change" is being assessed | 4 assessments will be carried out in the research in 10 weeks
  use of the affected upper extremity of spontaneous character during bimanual activities. It is used the AHA assessment to measure it.

SECONDARY OUTCOMES:
quality of life ,"change" is being assessed | 4 assessments will be carried out in the research in 10 weeks
  This measure will be assessed with the pedsQL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Palomo Carrión, Principal Investigator — Salamanca University
Locations (1):
- Rocío Palomo Carrión, Torrijos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tervahauta MH, Girolami GL, Oberg GK. Efficacy of constraint-induced movement therapy compared with bimanual intensive training in children with unilateral cerebral palsy: a systematic review. Clin Rehabil. 2017 Nov;31(11):1445-1456. doi: 10.1177/0269215517698834. Epub 2017 Mar 20. PMID 29050511
- [Result] Klepper SE, Clayton Krasinski D, Gilb MC, Khalil N. Comparing Unimanual and Bimanual Training in Upper Extremity Function in Children With Unilateral Cerebral Palsy. Pediatr Phys Ther. 2017 Oct;29(4):288-306. doi: 10.1097/PEP.0000000000000438. PMID 28953170
- [Result] Zafer H, Amjad I, Malik AN, Shaukat E. Effectiveness of Constraint induced movement therapy as compared to bimanual therapy in Upper motor function outcome in child with hemiplegic Cerebral palsy. Pak J Med Sci. 2016 Jan-Feb;32(1):181-4. doi: 10.12669/pjms.321.8491. PMID 27022371
- [Result] Geerdink Y, Aarts P, van der Burg J, Steenbergen B, Geurts A. Intensive upper limb intervention with self-management training is feasible and promising for older children and adolescents with unilateral cerebral palsy. Res Dev Disabil. 2015 Aug-Sep;43-44:97-105. doi: 10.1016/j.ridd.2015.06.013. Epub 2015 Jul 9. PMID 26164301
- [Result] Gelkop N, Burshtein DG, Lahav A, Brezner A, Al-Oraibi S, Ferre CL, Gordon AM. Efficacy of constraint-induced movement therapy and bimanual training in children with hemiplegic cerebral palsy in an educational setting. Phys Occup Ther Pediatr. 2015 Feb;35(1):24-39. doi: 10.3109/01942638.2014.925027. Epub 2014 Jul 1. PMID 24983295
- [Result] Sakzewski L, Gordon A, Eliasson AC. The state of the evidence for intensive upper limb therapy approaches for children with unilateral cerebral palsy. J Child Neurol. 2014 Aug;29(8):1077-90. doi: 10.1177/0883073814533150. Epub 2014 May 11. PMID 24820334
- [Derived] Palomo-Carrion R, Ferri-Morales A, Ando-LaFuente S, Fernandez RA, Arenillas JIC, Anton-Anton V, Esteban EB. Constraint-induced movement therapy versus bimanual intensive therapy in children with hemiplegia showing low/very low bimanual functional performance: A randomized clinical trial. PM R. 2023 Dec;15(12):1536-1546. doi: 10.1002/pmrj.12990. Epub 2023 Jun 19. PMID 37139775
- [Derived] Palomo-Carrion R, Lirio-Romero C, Ferri-Morales A, Jovellar-Isiegas P, Cortes-Vega MD, Romay-Barrero H. Combined intensive therapies at home in spastic unilateral cerebral palsy with high bimanual functional performance. What do they offer? A comparative randomised clinical trial. Ther Adv Chronic Dis. 2021 Aug 12;12:20406223211034996. doi: 10.1177/20406223211034996. eCollection 2021. PMID 34408823